CLINICAL TRIAL: NCT00998088
Title: Optimal Blood Management in Elective Orthopaedic Surgery: The Transfusion "Op Maat" (TOMaat) Study
Brief Title: Blood Management in Orthopedic Surgery
Acronym: TOMaat
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanquin Research & Blood Bank Divisions (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Roche BV Netherlands (Unknown); Haemonetics Corporation (Industry)
Responsible Party: Prof. Dr.R.G.H.H.Nelissen, Leiden University Medical Center
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: ISRCTN96327523; ISRCTN96327523; NTR303; ZonMW945-06-601; Sanquin PPOC-03-002
Record Dates: First submitted 2009-10-19; First posted 2009-10-20 (Estimated); Last update posted 2009-10-20 (Estimated); Status verified 2009-10

CONDITIONS: Osteoarthritis
Keywords: Blood management; Orthopedic surgery; elective; randomized study; adults; hip replacement; knee replacement
MeSH Terms: conditions — Osteoarthritis | interventions — Erythropoietin; Epoetin Alfa; epoetin beta; Drainage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Erythropoietin (Experimental)
  Interventions: Drug: erythropoietin
- Control arm (No Intervention)
- cell saver (Experimental)
  Interventions: Device: OrthoPAT
- drain (Experimental)
  Interventions: Device: Post-operative drain device
- Erythropoietin and cell saver (Experimental)
  Interventions: Other: erythropoietin and cell saver; Other: Erythropoietin and OrthoPAT
- Erythropoietin and drain (Experimental)
  Interventions: Other: Erythropoietin and drain device

INTERVENTIONS:
Other: erythropoietin and cell saver — weekly 40.000 IU s.c. for 4 weeks pre-operatively; use of cell saver includes intra- and post-operative drainage and reinfusion
  Other Names: Eprex, Ortho-Biotech; Neorecormon, Roche; OrthoPAT, Haemonetics
  Arms: Erythropoietin and cell saver
Drug: erythropoietin — weekly 40.000 IU s.c. for 4 weeks pre-operatively
  Other Names: Eprex, Ortho-Biotech; Neorecormon, Roche
  Arms: Erythropoietin
Device: OrthoPAT — for intra- and post-operative re-infusion of autologous wound blood
  Other Names: OrthoPAT, Haemonetics
  Arms: cell saver
Device: Post-operative drain device — For post-operative re-infusion of unwashed wound blood
  Other Names: Bellovac-ABT, Astra-Tech, The Netherlands; DONOR-drain, Van Straten Medical, The Netherlands
  Arms: drain
Other: Erythropoietin and OrthoPAT — weekly 40.000 IU s.c. for 4 weeks pre-operatively
  Other Names: Eprex, Ortho-Biotech; Neorecormon, Roche; OrthoPAT, Haemonetics
  Arms: Erythropoietin and cell saver
Other: Erythropoietin and drain device — weekly 40.000 IE s.c.for 4 weeks pre-operatively; drain use in post-operative period
  Other Names: Eprex, Ortho-Biotech; Neorecormon, Roche; Bellovac-ABT, Astra-Tech; DONOR-drain, Van Straten Medical
  Arms: Erythropoietin and drain
Device: OrthoPAT — For intra- and post-operative reinfusion of autologous blood
  Other Names: OrthoPAT, Haemonetics
  Arms: cell saver

SUMMARY:
Aim: to investigate whether the use of several transfusion alternatives (erythropoietin, the cell-saver or postoperative drainage and reinfusion systems) in patients undergoing elective total knee or hip replacement surgery can lead to allogeneic red blood cell (RBC) saving if a restrictive transfusion policy is used.

Study design: a prospective, double randomized, open, multicenter study in which patients are stratified according to their preoperative hemoglobin(Hb) level: stratum I= Hb between 6,1 and 8,2 mmol/l. These patients are first randomized for Erythropoetin (Epo) or no Epo.

Stratum II= Hb of 6,1 and lower or 8,2 mmol/l and higher, are not eligible for Epo and thus not randomized. Patients in both strata will be randomized for three modalities: a cell saver (CS)(to wash, filter and reinfuse autologous shed blood) which is used intra- and postoperatively or a postoperative autologous reinfusion drainage system (D) only (to filter and reinfuse autologous shed blood) or a restrictive transfusion trigger only (controls).

Inclusion criteria: All orthopedic patients of 18 years and older being considered for a primary or revision total knee- (TKR) or total hip replacement (THR).

Outcome measures:

Primary outcome: number of allogeneic red blood cell (RBC) transfusions.

Secondary outcome: transfusion reactions, rehabilitation time, length of hospital stay (days), peri- and post-operative complications during hospitalization, quality of life, cost analysis

DETAILED DESCRIPTION:
Power/data analysis: In order to be able to detect a 75% reduction of allogeneic transfusions by Epo and a reduction of 30% by autologous (shed blood) transfusions (CS or D) with a power= 0.9 and an alpha= 0.05, inclusion of 2250 surgery patients (in a worst case scenario of high standard deviations) are required for intention-to-treat analysis.

Knee surgery patients are not randomized for cell saver (no intra-operative blood loss).

ELIGIBILITY:
Inclusion Criteria:

* Orthopaedic patients of 18 years and older being scheduled for a primary or revision total knee (TKR) or total hip replacement (THR).

Exclusion Criteria:

* Patients who refuse homologous blood (e.g.Jehovah's witnesses),
* Patients with untreated hypertension (diastolic blood pressure > 95 mm Hg),
* Patients with a serious disorder of the coronary artery, peripheral arteries and/or carotid arteries,
* A recent myocardial infarction or CVA,
* Sickle cell anaemia patients,
* Malignancy in the operated area,
* Pregnancy,
* Unsuitability for peri-operative anticoagulation prophylaxis,
* Known allergy to erythropoietin,
* An infected wound bed,
* Revision of an infected prosthesis which is being treated with antibiotics, OR
* Patients with difficulty understanding the Dutch language (unable to give informed consent or patients who insufficiently control the Dutch language).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2598 (Actual)
Dates: Start 2004-05; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Number of allogeneic red blood cell (RBC) transfusions. | up to 3 months after surgery

SECONDARY OUTCOMES:
Peri- and post-operative complications during hospitalization | up to 3 months after surgery
Rehabilitation time | in hospital
Hb/Ht post-operative | at 14 days and 3 months after surgery
Quality of life | Up to 3 months after surgery
Transfusion reactions | up to 3 months after surgery
Harris hip / knee society score (for determination of the mobility of the operated joint) | pre-operative and after 3 months
Cost analysis | up to 3 months after surgery
Length of hospital stay | In hospital

CONTACTS AND LOCATIONS:
Overall Officials: Rob Nelissen, MD, PhD, Principal Investigator — Leiden University Medical Center
Locations (4):
- Netherlands (4):
  - Slotervaart Hospital, Amsterdam, North Holland
  - Albert Schweitzer Hospital, Dordrecht, South Holland
  - Groene Hart Hospital, Gouda, South Holland
  - LUMC, Leiden, South Holland